CLINICAL TRIAL: NCT00378638
Title: Dose-Dense Chemotherapy Plus Bevacizumab in High Risk Lymp Node Positive Breast Cancer: A Pilot Study
Brief Title: Dose-Dense Chemotherapy Plus Bevacizumab in High Risk Lymph Node Positive Breast Cancer: A Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chap, Linnea I., M.D. (Individual)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3359s; NCT00372866 (obsolete NCT alias)
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2007-10-24 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: lymph; node; positive; breast; cancer; metastases; angiogenesis; bevacizumab; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bevacizumab combined with dose dense chemotherapy

SUMMARY:
This research focuses on women with breast cancer whose disease has not significantly progressed, but who have 5 or more lymph nodes involved. In this study subjects will receive bevacizumab, a drug which is FDA approved for colon cancer but not for breast cancer, in combination with a regimen of approved chemotherapy drugs known as "dose dense chemotherapy." The study will observe the effectiveness and tolerability of this regimen.

DETAILED DESCRIPTION:
Approximately 200,000 women are diagnosed with breast cancer in the United States every year. A significant factor determining long-term survivability of breast cancer is whether or not lymph nodes, glands which cleanse and filter the body's fluids, are involved. Despite treatment with approved multiagent cytotoxic chemotherapy ("dose-dense chemotherapy"), women with breast cancer involving more than 4 axillary lymph nodes still have a high risk for recurrence.

Several dose-dense chemotherapy regimens are currently being compared in other studies, however, at this time there is no proof that one regimen is superior to another. Therefore, in an attempt to decrease metastases, prolong time to recurrence and improve overall survival, it is essential to develop novel therapeutic strategies. The use of inhibitors of angiogenesis represents a promising option.

Bevacizumab is the first angiogenesis inhibiting drug to be FDA approved, for the treatment of colon cancer. It is has also been studied alone in progressed lymph-node positive breast cancer and has shown moderate efficacy.

This study will observe the efficacy and tolerability of using bevacizumab in combination with an approved dose-dense chemotherapy regimen for 8 cycles, followed by 12 of bevacizumab alone. Patients may be on the study for up to 52 weeks if their disease has not progressed and the regimen is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* High risk lymph node positive breast cancer defined as 5 or more involved axillary lymph nodes
* Must have undergone surgical local therapy (modified radical mastectomy or breast conserving surgery).
* Negative tumor margins for invasive cancer
* No evidence of distant metastasis
* Normal cardiac ejection fraction
* Adequate organ function defined as:

ANC > 1200/mm3 Platelet count > 100,000/mm Serum creatinine < 2.0 mg/dl Serum bilirubin < 1.5 x ULN

* Performance status 0-1
* Age 18 years or older
* No prior chemotherapy, hormonal therapy or radiation therapy for treatment of the primary breast cancer
* Bilateral synchronous breast cancer is allowed if other criteria are met.
* Patients may be ER/PR+ and receive treatment with hormonal therapy (tamoxifen or aromatase inhibitors)
* Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Signed informed consent

Exclusion Criteria:

* Evidence of distant metastases
* Inflammatory Breast Cancer
* Prior use of any chemotherapy or hormonal therapy for breast cancer
* Patients with her 2 neu positive tumors
* History of other malignancies within the last 5 years. Prior history of carcinoma in situ of the cervix, melanoma in situ and basal cell carcinoma of the skin is allowed within the last 5 years.
* Prior therapy with anthracyclines for any malignancy
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Blood pressure of equal to or higher than 150/100
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein:creatinine ratio >1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-06; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment failure, 2 and 5 year Disease Free Survival.

SECONDARY OUTCOMES:
2 and 5 Year Disease Free Survival.
Overall survival.
Circulating Tumor Cells and Circulating Endothelial Progenitor Cells assays results and their association with clinical outcomes.
Toxicities and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Linnea I. Chap, MD, Principal Investigator — Premiere Oncology, A Medical Corporation
Locations (1):
- Premiere Oncology, Santa Monica, California, United States